CLINICAL TRIAL: NCT01050270
Title: A Randomised Trial to Assess the Effectiveness of Pre-treatment With Ondansetron at Reducing Nausea and Vomiting in Patients Treated With Either the Conventional Regimen or a Modified Regimen of Acetylcysteine for Paracetamol Poisoning
Brief Title: Scottish and Newcastle Anti-emetic Pre-treatment for Paracetamol Poisoning Study (SNAP)
Acronym: SNAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZB/4/722; 2009-017800-10 (EudraCT Number)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Overdose
MeSH Terms: conditions — Drug Overdose | interventions — Ondansetron; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ondansetron /acetylcysteine 20.25h (Other): Ondansetron followed by conventional acetylcysteine regimen
  Interventions: Drug: Ondansetron; Drug: acetylcysteine
- Placebo/acetylcysteine 20.25h (Other): placebo followed by conventional acetylcysteine regimen
  Interventions: Drug: acetylcysteine
- Ondansetron/acetylcysteine 12h (Other): ondansetron followed by modified acetylcysteine regimen
  Interventions: Drug: Ondansetron; Drug: acetylcysteine
- Placebo/acetylcysteine 12h (Other): placebo followed by modified acetylcysteine regimen
  Interventions: Drug: acetylcysteine

INTERVENTIONS:
Drug: Ondansetron — 4mgs iv bolus
  Other Names: CAS number: 99614-02-5
  Arms: Ondansetron /acetylcysteine 20.25h; Ondansetron/acetylcysteine 12h
Drug: acetylcysteine — 100 mg/kg over 2 hours then 200mg/kg over 10 hours, followed by glucose 5% for 8 hours
  Other Names: cas number: 616-91-1
  Arms: Ondansetron/acetylcysteine 12h; Placebo/acetylcysteine 12h
Drug: acetylcysteine — 150 mg/kg over 15 mins 50 mg/kg over 4 hours 100 mg/kg over 16 hours
  Other Names: CAS number: 616-91-1
  Arms: Ondansetron /acetylcysteine 20.25h; Placebo/acetylcysteine 20.25h

SUMMARY:
This study is designed to assess the impact of new approaches to therapy for paracetamol poisoning. Standard therapy is currently acetylcysteine by intravenous infusion over 20.25h. This regimen is given to those deemed "at risk" using standard criteria (British National Formulary 200920). It has 3 major problems, adverse events (nausea and vomiting and anaphylactoid reactions), therapy duration and complexity of administration.

This study is primarily designed to test the efficacy of prophylactic anti-emetic therapy.

It will also provide sufficient experience and data from a modified shortened IV acetylcysteine regimen to adequately design and power a study of the modified regimen as a new treatment for this common poison. Such an approach has a major potential to reduce patient adverse events from acetylcysteine therapy and shorten duration of hospital stay.

DETAILED DESCRIPTION:
Paracetamol is the commonest poison seen in the United Kingdom and is present in approximately 40% of patients admitted with self harm. Current treatment involves use of the antidote acetylcysteine in patients deemed at risk of potential liver damage. This is given by intravenous infusion over a period of 20.25 hours. This regimen was designed in the 1970s and is empirical, in that a large loading dose of the antidote is administered followed by 2 decreasing concentrations. It is cumbersome to calculate and dilute within the ward and therefore subject to error in preparation. The initial infusion is associated with a significant rate of adverse reactions, in particular nausea and vomiting and anaphylactoid reactions. The latter are particularly troublesome and occur in up to 15% of patients treated. Therapy is discontinued and there is often confusion as to whether it can be restarted in a timely manner.

Studying antidotes in the management of poisoning is challenging not least because of the patient population and of the limited time available to make decisions and gain consent. This will be the first major clinical trial of antidote therapy in this poisoning in the UK in 30 years.

The final objective of this work is to develop a therapeutic regimen of acetylcysteine that does not cause such a high rate of adverse reactions and is also easier for nurses to make up.

The present study focuses on the potential use of ondansetron, an anti-emetic, prior to the administration of acetylcysteine. It will also allow preliminary data to be collected on a new approach to giving acetylcysteine using a modified 12 h regimen, which includes a slower initial intravenous infusion.

The primary trial outcome will therefore inform on the efficacy of ondansetron pre-treatment as an anti-emetic in this situation. In addition valuable data on the incidence of adverse effects caused by the modified acetylcysteine regimen, and changes in liver function and the inflammatory response to paracetamol liver injury caused by paracetamol within this modified acetylcysteine treatment will be obtained.

In addition an opportunity will be taken in a convenience sample of 40 patients to study the pharmacokinetics of acetylcysteine in this group using the standard and modified regimens.

A factorial design is being used to answer the key clinical questions. In total a maximum of 250 patients will be recruited and it is anticipated the data from 200 will be available for final analysis.

The demographic of this patient group is essentially Caucasian English-speaking and at this stage we do not propose to recruit non-English-speaking subjects.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to hospital within 36 hours of a single acute paracetamol overdose; AND
* Requires treatment with acetylcysteine.

These patients will include:

* Patients with no risk factors and timed paracetamol concentrations above the 200-line on the UK paracetamol overdose treatment nomogram.
* Patients with at least 1 risk factor and timed paracetamol concentrations above the 100-line on the UK paracetamol overdose treatment nomogram
* Patients presenting >8 hours, and at risk of liver damage based on history of dose ingested (BNF) that need immediate treatment

Risk factors are defined as follows:

* Nutritional deficiency, malnourished and/or debilitating disease: acute or chronic starvation, eating disorders, cachexia, malabsorption syndromes, AIDS, cystic fibrosis, hepatitis C, chronic alcoholism.
* Enzyme induction: use of drugs with this property (carbamazepine, rifampicin, barbiturates, phenytoin, rifabutin, efavirenz, nevirapine, St John's Wort; regular consumption of ethanol above advised amounts.

Exclusion Criteria:

Patients:

* < 16 years old
* Detained under the Mental Health Act
* With known permanent cognitive impairment
* With a life-threatening illness
* Who are known to be pregnant
* Who have previously participated in the study
* Unreliable history of paracetamol overdose
* Vomiting and requiring treatment antiemetic prior to randomisation
* Presenting after 36 hours of a single acute paracetamol overdose
* Presenting after taking a staggered paracetamol overdose (defined as when the overdose of paracetamol is taken over a period of more than 2 hours)
* Who take anticoagulants (e.g. warfarin) therapeutically or have taken an overdose of anticoagulants
* Who, in the opinion of the responsible clinician/nurse, are unlikely to complete the full course of acetylcysteine e.g. expressing wish to self-discharge
* Who in the opinion of the responsible clinician/nurse are unable to complete the initial questionnaire either themselves or with nurse assistance.
* Who have a history of hypersensitivity to 5HT3 antagonists
* Non-English speaking patients. (Trial information material will only be produced in English in view of the known and stable demographic of the Edinburgh and Newcastle self harm population)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of patients who do not vomit or retch within 2 hours of initiation of acetylcysteine treatment and no use of rescue medication. Retching will be defined as a vomit not producing any liquid. | 2 hours post start of treatment

SECONDARY OUTCOMES:
The secondary endpoint is nausea or vomiting within 12h of initiation of acetylcysteine treatment. | 12 hours post start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair J Gray, Principal Investigator — NHS Lothian; Harry K Thanacoody, Principal Investigator — Newcastle Hospitals NHS Foundation Trust; Jamie G Cooper, Principal Investigator — NHS Grampian
Locations (3):
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Derived] Bateman DN, Dear JW, Thanacoody HK, Thomas SH, Eddleston M, Sandilands EA, Coyle J, Cooper JG, Rodriguez A, Butcher I, Lewis SC, Vliegenthart AD, Veiraiah A, Webb DJ, Gray A. Reduction of adverse effects from intravenous acetylcysteine treatment for paracetamol poisoning: a randomised controlled trial. Lancet. 2014 Feb 22;383(9918):697-704. doi: 10.1016/S0140-6736(13)62062-0. Epub 2013 Nov 28. PMID 24290406
- [Derived] Thanacoody HK, Gray A, Dear JW, Coyle J, Sandilands EA, Webb DJ, Lewis S, Eddleston M, Thomas SH, Bateman DN. Scottish and Newcastle antiemetic pre-treatment for paracetamol poisoning study (SNAP). BMC Pharmacol Toxicol. 2013 Apr 4;14:20. doi: 10.1186/2050-6511-14-20. PMID 23556549